CLINICAL TRIAL: NCT04155242
Title: Prospective Study on the Use of Biomarkers to Guide Management of Patients Treated With Radiofrequency Ablation for Early Oesophageal Neoplasia
Brief Title: The Use of Biomarkers to Guide Management of Patients Treated With Radiofrequency Ablation for Early Oesophageal Neoplasia
Acronym: PROBAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, Massimiliano di Pietro, MD, Dr Massimiliano di Pietro, Senior Clinical Investigator Scientist, MRC Cancer Unit, Hutchison-MRC Research Hon. Consultant Gastroenterologist, Addenbrooke's Hospital, Cambridge., University of Cambridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISRCTN12730505
Record Dates: First submitted 2019-10-25; First posted 2019-11-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Barrett's Oesophagus
Keywords: Barrett's oesophagus; Radiofrequency ablation; Early Oesophageal Neoplasia
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): As part of the post RFA treatment follow up patients will receive a Cytosponge test followed by an endoscopy with NBI magnification and biopsies. Four endoscopies will be performed during 2 years of active follow up together with up to 2 Cytosponge procedures. Molecular biomarkers including a methylation panel on DNA and immunohistochemical markers on formalin fixed paraffin embedded samples obtained during the examinations will be assessed. Patients will be then followed up for up to 3 years with standard endoscopy to assess for relapse of Barrett's oesophagus/IM/dysplasia.
  Interventions: Diagnostic Test: Cytosponge test; Diagnostic Test: Assessment of the panel of molecular biomarkers: IM-SCORE, TFF3 protein expression, methylation panel, p53 mutation; Diagnostic Test: Oesophagogastroduodenoscopy

INTERVENTIONS:
Diagnostic Test: Cytosponge test — The Cytosponge will be administered by the study nurse prior to the participant having the endoscopy, usually as part of the same visit to hospital. The capsule along with the string is swallowed by drinking a small glass of water. The participant is asked to hold the Cytosponge in situ for 5 minutes. The sponge contained within expands and is then drawn back by the research nurse up the oesophagus by the attached string, collecting cells as it moves upwards. This device received a letter of no objection by the MHRA for use in the BEST pilot trial (LRQ 0939857) but it is not CE marked. Cytosponge and research endoscopic biopsies will be couriered to the Fitzgerald laboratory, at the MRC Cancer Cell Unit on a regular basis. The specimens will be processed in conjunction with the Cambridge University Hospitals' NHS Foundation Trust tissue bank which is accredited to GLP standards.
Diagnostic Test: Assessment of the panel of molecular biomarkers: IM-SCORE, TFF3 protein expression, methylation panel, p53 mutation — Molecular analysis of the specimen obtained by Cytosponge or endoscopic biopsies - TFF3 protein expression, methylation panel, p53 mutation. Endoscopic biopsies will be assessed for the presence of IM (according to the IM-score).
Diagnostic Test: Oesophagogastroduodenoscopy — * Endoscopy will be carried out with white light and NBI with optical magnification or near focus to inspect oesophagus and GOJ.
  * NBI magnification will be used to assess systematically the mucosal pit pattern at the GOJ and to look for light blue crest (LBC) sign.
  * Targeted biopsies will be taken from either areas with LBC or irregular pit pattern on NBI, followed by random biopsies as per clinical standard. A maximum of 6 biopsies will be taken at the GOJ (maximum 4 targeted and 4 random.. During the first 2 post RFA follow up, at discretion of the endoscopists, neo-suqamous biopsies can be taken in line with local policies.
  * Argon plasma coagulation ablation is allowed in a single island up to 5mm or up to 3 islands <3mm within the study endoscopy as long as this does not represent an obstacle to GOJ biopsies.

SUMMARY:
This prospective cohort study aims to assess the utility of a panel of molecular biomarkers for predicting the risk of relapse of Barrett's Oesophagus after endoscopic treatment of early oesophageal neoplasia with RadioFrequency Ablation (RFA). Patients who received endoscopic treatment of early oesophageal neoplasia with RFA and achieved endoscopic remission will be recruited. During the surveillance visits patients will receive a Cytosponge test followed by an endoscopy with Narrow Band Imaging (NBI) magnification and biopsies. Patients will receive an endoscopy every 6 months and Cytosponge every 12 months for at least 2 years. Molecular biomarkers including a methylation panel on DNA and immunohistochemical markers on formalin fixed paraffin embedded samples. After 2 years of intensive endoscopic follow up, patients will be prospectively tracked for up to 3 years.

The investigators will also evaluate:

* The risk of progression to dysplasia or oesophageal intestinal metaplasia (IM) in patients with IM at the GOJ post RFA in the absence of retreatment
* the diagnostic accuracy of NBI for IM/dysplasia at the GOJ .

DETAILED DESCRIPTION:
The panel of predetermined molecular biomarkers includes:

1. IM-SCORE - a score quantifying the extent of intestinal metaplasia at GOJ, which uses a 4-tier system based on the number of glands and the number of biopsies with features of IM. The score has been developed in a pilot study (manuscript under submission) and will be validated in this study
2. Methylation markers- assessed by a PCR-based method (Methylight) on Cytosponge samples.
3. P53 status.
4. TFF3 protein expression.

ELIGIBILITY:
Inclusion Criteria

1. Previous RFA for dysplastic BE or following EMR for BE-related neoplasia
2. No definite endoscopic evidence of BE defined as at least 1cm tongue of columnar oesophagus or oesophageal BE islands larger than 5mm.
3. No histological evidence of oesophageal IM including buried BE at first post RFA follow up. GOJ IM is allowed
4. No evidence of suspicious lesions with dysplasia at the GOJ.

Exclusion criteria

1. Evidence of BE requiring additional RFA
2. Anticoagulant or antiplatelet therapy for high risk conditions, whereby discontinuation of the treatment is not recommended.
3. Individuals with a diagnosis of an oro-pharynx, oesophageal or gastro-oesophageal tumour (T2 staging and above), or symptoms of dysphagia,
4. Oesophageal varices, stricture or requiring dilatation of the oesophagus
5. Individuals who have had a myocardial infarction or any cardiac event less than six months ago
6. Patients whose primary previous ablative treatment was different from RFA, such as Photodynamic therapy (PDT), APC or Cryotherapy
7. Participants who are unable to provide informed consent.
8. Participants under age 18.
9. Endoscopy is generally avoided in pregnant women and therefore it is unlikely that any pregnant women will be included although pregnancy would not be an absolute contraindication. Pregnancy/ pregnancy test will not be recorded as part of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of methylation panel for diffuse IM at the GOJ | 5 years
  Diagnostic accuracy of a panel of methylation markers (ZNF345, ZNF569 and TFPI2 loci) for diffuse IM at the GOJ assessed by Methylight on DNA extracted from GOJ biopsies (separately random and targeted biopsies) and Cytosponge samples.

SECONDARY OUTCOMES:
Proportion of patients developing true BE recurrence | 5 years
  Number of patients with GOJ IM with different IM score that will develop true BE recurrence during the observation period defined as oesophageal IM or dysplasia.
Biomarker score for BE recurrence | 5 years
  The accuracy of a biomarker panel to predict risk of BE recurrence. The following biomarkers will be assessed:
  * P53 status by immunohistochemistry
  * TFF3 expression by immunohistochemistry
  * IM-SCORE (defined in the Study Description section)
  * methylation markers (defined in the Outcome 1 Description section).
Accuracy of Light Blue Crest sign | 5 years
  Diagnostic accuracy of a Light Blue Crest (LBC) sign in NBI for the diagnosis of GOJ IM. During each performed endoscopy, NBI magnification will be used to assess systematically the mucosal pit pattern at the GOJ and to look for the LBC sign. In order to assess the accuracy of LBC, targeted biopsies will be taken from all the areas with LBC.
Safety of Cytosponge | 5 years
  Number of participants with Cytosponge procedure-related serious adverse events defined as an event that:
  Results in death Is life-threatening Requires hospitalisation or prolongation of existing hospitalisation Results in persistent or significant disability or incapacity Consists of a congenital anomaly or birth defect Is otherwise considered medically significant by the investigator (eg. a further procedure is required for the patient).

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Di Pietro, MD, Principal Investigator — MRC Cancer Unit, Hutchison-MRC Research Hon. Consultant Gastroenterologist, Addenbrooke's Hospital, Cambridge.
Locations (1):
- MRC Cancer Unit, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No